CLINICAL TRIAL: NCT02353338
Title: Distal Radial Fractures in the Late Middle Aged: Surgical or Conservative Treatment - A Randomized Control Trial
Brief Title: Distal Radial Fractures in the Late Middle Aged
Acronym: RIST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RES0025250
Record Dates: First submitted 2015-01-28; First posted 2015-02-02 (Estimated); Last update posted 2021-09-22 (Actual); Status verified 2021-09

CONDITIONS: Radius Fracture
MeSH Terms: conditions — Radius Fractures | interventions — Surgical Procedures, Operative; Conservative Treatment; Casts, Surgical

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A: Surgical (Experimental): Individuals in Group A will receive surgery to correct their radial fracture
  Interventions: Procedure: Surgical intervention
- Group B: Conservative Treatment (Active Comparator): Individuals in Group B will be immobilized in a cast, as per usual standard of conservative treatment.
  Interventions: Procedure: Conservative management; Device: cast

INTERVENTIONS:
Procedure: Surgical intervention — Surgical management of radial fracture
  Arms: Group A: Surgical
Procedure: Conservative management — Immobilized/cast for 6 weeks
  Arms: Group B: Conservative Treatment
Device: cast
  Arms: Group B: Conservative Treatment

SUMMARY:
Background: Wrist fractures are a common injury among people aged 55-70. The radius is one of the bones making up the wrist joint, and is typically the site of injury in a broken wrist. Methods of treating a broken radius include placing the wrist in a cast for 6 weeks (conservative management) or receiving surgery. Surgery allows for earlier movement of the wrist and return to activity, while being placed in a cast is less invasive than surgery.

Surgery to fix these fractures has become more common; however there is little agreement about who should receive surgery and who should be placed in a cast to heal. The goal of this study is to compare outcomes between people aged 55-70 who have broken their wrist and had surgery, and those who received a cast.

Procedures: Participants in this study will be randomly assigned to one of two study groups within 1 week of injury at their first clinic visit with the surgeon.

Patients in Group A (surgical management) will continue with casting for a total of 6 weeks, as indicated by the surgeon.

Patients in Group B (conservative management) will receive surgery, and the attending surgeon will determine the best fracture fixation method for the wrist.

The research coordinator will assess the injured wrist at 6 weeks, 3, 6, and 12 months after the initial injury. At each assessment, the wrist will be examined and participants will be asked to fill in some questionnaires about health, pain, wrist function, and satisfaction with the wrist. An X-ray will also be performed on the wrist to assess bone healing. Information from each visit will be used to determine how participants are doing and to compare the 2 study groups.

DETAILED DESCRIPTION:
BACKGROUND

Distal radius fractures (DRF) are the most common upper extremity fractures in late middle-aged patients. This injury creates significant disability rendering a person without full use of the affected hand and wrist for 6 weeks or more with potential long-term consequences of post-traumatic wrist arthritis and contracture. Over the past 20 years, surgical management of DRF has increased substantially. Despite the frequency of these fractures, there is little comparative evidence to guide surgical decision-making for this population.

Although surgical management improves radiographic outcomes, it does not appear that radiographic outcomes correlate well with patient reported outcomes (pain and function). As there are significant health resource implications of surgical versus conservative management, it is imperative that we determine when operative fixation is needed. Further, as our population is aging, the number of patients with DRF will increase substantially in the late to middle-aged and elderly adults.

For subjects under 55 years of age, surgical management is often undertaken to allow early mobility and facilitate return to work and activity, even in the presence of equivocal clinical outcomes between management approaches. Conversely, in those who are older than 70 years, conservative management is more common due to lower patient demands.

However, the American Academy of Orthopedic Surgeons issued clinical practice guidelines that could not make evidence based treatment recommendations for patients aged 55 to 70 years with DRFs. Thus, there is no current available evidence comparing patient outcomes between surgical and conservative management in this age group. The overall goal of RIST will be to compare outcomes between patients aged 55-70 years who receive surgical or conservative management. Our primary outcome will be a clinical measure (patient-reported or performance-based) rather than radiographic alignment.

Because evidence focused around this age group is sparse, we will first conduct a pilot trial to clarify eligibility criteria, outcome measure selection, sample size requirements, and recruitment and retention rates. In 2013, 610 patients aged 55-70 years with DRFs were seen in Edmonton emergency departments and 314 inpatients aged 55-70 years with DRFs were discharged from all hospitals in the greater Edmonton area.

OBJECTIVES

Primary objective: To determine the feasibility of conducting a definitive RCT comparing surgical versus conservative management in 55-70 year old patients with DRF. This study will examine:

1. Recruitment and eligibility rates
2. Treatment fidelity (the ability to deliver the intervention in the way that it was intended) through measurement of patient crossovers from non-operative management to operative fixation within the first year of fracture
3. Outcomes and outcome measures to determine most appropriate measure and sample size required
4. Retention rate at 1 year.

Secondary objective: To compare clinical and radiographic outcomes of surgical and conservative management for 55-70 year old patients with DRF over the first year post-fracture using:

1. Patient-Rated Wrist Evaluation (PRWE) Questionnaire - currently deemed primary outcome measure
2. Disabilities of the Arm, Shoulder and Hand (DASH) Questionnaire
3. Patient satisfaction regarding cosmesis using a visual analogue scale (VAS)
4. Grip strength using a hand-held dynamometer
5. Wrist Range of Motion (ROM) using standardized goniometry
6. Radiographic measures (dorsal angulation, ulnar shortening, articular steps and gaps.)

EXPERIMENTAL PROTOCOL

Study Design: Parallel RCT with stratification by surgeon using computer generated unequal randomization blocks. Following screening, consent and baseline evaluation, the research coordinator will open sequentially numbered envelopes assigned to the treating surgeon. Participants will be randomized to operative fixation or cast treatment.

Selection Criteria: This pilot RCT will enroll 55 to 70 year old subjects with isolated intra- or extra-articular displaced DRFs who present to the Sturgeon Community Hospital (SCH) for medical care under 1 of 5 fellowship-trained upper-extremity orthopaedic surgeons. Eligible subjects will present with the following radiographic findings before reduction: dorsal angulation ≤20 degrees, ulnar shortening ≤5 mm relative to the contralateral side (subjects will have contralateral wrist xrays), articular step ≤2 mm after initial post reduction and gap ≤5 mm. These parameters were chosen as they meet accepted criteria for distal radius fracture instability, but are still correctable by osteotomy if the fracture heals with this degree of mal-alignment.

Patients with volar Barton fractures, radiocarpal subluxation or dislocation, open fractures, ipsilateral upper extremity injuries, bilateral fractures or multiple traumas will be excluded. Those with previous injury or fracture to the contralateral wrist, or those not fit for surgical management will also be excluded.

Screening and Enrollment: Patients will be screened for study eligibility at their initial clinic visit by the attending surgeon and research coordinator within 1 week of injury. The Research Coordinator will track reasons for refusal from patients who do not consent to participate as well as exclusions by the surgeons based on patient or fracture characteristics. Those patients who agree to participate will be consented and enrolled by the Research Coordinator. The baseline evaluation will consist of completion of a demographics/screening form form (age, gender, mechanism of injury, past and current medical status, work and activity demands) and PRWE and DASH questionnaires. All data will be collected using standardized forms and entered into a password-protected database.

Intervention: Following the baseline evaluation, the subject will be randomized to receive either surgical or conservative management. Those with conservative management will continue with casting for a total of 6 weeks. For those randomized to operative fixation, the attending surgeon will determine the optimal fracture fixation method for the fracture pattern.

At each follow-up visit, the surgeon, in conjunction with the patient, will evaluate outcomes in the conservatively managed group to determine if corrective osteotomy is indicated based on the patient's pain, weakness and acceptance of clinical deformity. If a corrective osteotomy is required at any time point in the study, this will be considered as failure of non-operative treatment. This approach is being used in the feasibility trial to assess the current selection criteria to determine if they require revision prior to the definitive RCT.

Follow-up Evaluations: Two weeks after randomization, the research coordinator will contact participants by telephone to complete the PRWE and Dash questionnaires, and ask about any complications related to their injury. Participants will return to clinical follow-up at 6 weeks, 3 months, 6 months and 12 months at the SCH using the same validated measures. Starting at the 6 week assessment, wrist ROM (flexion, extension, pronation, supination, ulnar and radial deviation) using a goniometer and grip strength using a hand-held dynamometer will also be evaluated by the research coordinator. Radiographic evaluation of dorsal angulation, ulnar shortening, articular steps and gaps and complications and adverse events will also be recorded at each visit. At 1-year follow-up, patient satisfaction with their clinical outcome will be assessed using a PRWE and DASH questionnaires and a VAS for determining satisfaction with wrist cosmesis.

Outcomes and Outcome Measures: Although radiographic parameters will be collected and measured, the primary outcomes will be the clinical measures: patient-reported wrist specific outcomes (PRWE), patient reported upper extremity function (DASH) and wrist ROM and grip strength.

1. Patient-Rated Wrist Evaluation (PRWE) Questionnaire - The PRWE is a brief, reliable and valid 15-item tool used to assess patient-rated wrist pain and disability during activities of daily living. Subjects rate their pain and function from 0-10 in two different subscales: pain subscale and function subscale. The minimally clinically important difference (MCID) for the PRWE is 17 points on a 0-100 score.
2. Disabilities of the Arm, Shoulder and Hand (DASH) Questionnaire - The DASH is a valid and reliable 30-item scale that assess physical function and symptoms in subjects with upper limb musculoskeletal issues. It has three modules: disability and symptom (mandatory), work (optional) and sports/performing arts (optional). The MCID for the DASH is 13 points on a 0-100 score.
3. Patient satisfaction - Patient satisfaction with their outcome is in part being answered with the PRWE and DASH questionnaires, since both assess pain and function. However, because we are comparing surgical versus conservative treatment, it is also important to evaluate how satisfied the subjects are with the cosmesis of their wrist after treatment. Conservative treatment may leave a mal-aligned wrist and surgical treatment will leave scars and the acceptability of either may affect the willingness of the subject to agree with either treatment choice. Therefore, we will use a visual analogue scale to measure how satisfied the subject is with the cosmesis of the wrist after treatment (0- not satisfied at all to 10- completely satisfied).
4. Grip strength - Peak values of grip strength in both hands will be measured with a hand-held dynamometer. Absolute values and percentage of their contralateral side will be compared between the two groups. The MCID for grip strength after DRF is 6.5 kilograms or 20%.
5. Wrist Range of Motion (ROM) - Active and passive ROM of wrist flexion, extension, ulnar deviation, radial deviation, pronation and supination will be assessed using goniometry. Absolute values and percentage of their contralateral side will be compared between groups. No MCID have been established for wrist ROM, so we will evaluate differences in ROM and correlate those with both grip strength and patient reported outcomes to determine what differences in ROM appear to affect outcomes, if any.
6. Radiographic Parameters: Dorsal angulation, ulnar shortening, articular steps and gaps will be measured at initial presentation and when fracture is healed (6 weeks) and at the end of the study period (12 months).

Sample Size: For this feasibility trial, 50 participants (25/group) will be enrolled. This will allow us to assess subject recruitment, treatment fidelity and retention. Based on our findings, we will refine our selection criteria as necessary for the definitive RCT. This pilot evaluation will provide for calculation of the sample size for the definitive RCT based on confirmation of the primary outcome measure. Although 50 participants will likely be inadequate to detect significant group differences, it should be adequate to determine if MCID occur in clinical outcomes between groups.

Analysis: The analysis of this feasibility component of the RIST trial will be 2-pronged to prepare for the definitive RCT:

1. Process Evaluation: This process evaluation will be a descriptive analysis that will assist us in refining eligibility criteria, recruitment rates, treatment fidelity and determine study timelines prior to undertaking a large scale RCT.

   Recruitment, enrollment and retention rates: All 55-70 year old DRF patients presenting at the SCH will be screened so that eligibility, recruitment and retention rates can be assessed. We will also evaluate recruitment methods to determine the proportion of patients 1) willing to participate and 2) appropriate for randomization.
2. Treatment Fidelity: We will assess failure of allocation to treatment by examining the numbers of patients that withdraw post randomization or cross over to surgical management within the first post-fracture year. This will determine if selection criteria require further refinement.

Intervention Evaluation: Our secondary objective is to compare outcomes between randomized groups. T-tests and repeated measures analysis of variance (ANOVA) will be used with continuous variables and chi square tests will be performed on categorical variables.

Outcome Selection: We believe that the PRWE will be the most responsive measure as it is patient-reported wrist specific pain and function. However, we will also evaluate the DASH, cosmesis satisfaction (VAS) and the performance-based measures of grip strength and wrist ROM. Radiographic parameters will not be considered as primary outcomes because previous work has suggested the clinical and radiographic parameters are not well-correlated in DRF.

Sample Size Calculation: The intervention analysis will also allow us to determine if we should perform a superiority or inferiority RCT. If there are no MCID detected in the pilot study (expected), the definitive RCT will be powered as a non-inferiority trial (i.e. similar clinical outcomes can be achieved with surgical or conservative management in this age group). If MCID are found in clinical measures, the definitive RCT will be powered as a superiority trial (e.g. surgical fixation is better than conservative treatment).

Expected Outcome: This proposed pilot study is important for assessing the feasibility of conducting a definitive RCT so that potential challenges can be addressed prior to commencing the larger-scale trial. The pilot data generated will be used to develop a grant proposal for an adequately-powered definitive RCT. However, we believe that the pilot study will be appropriate for presentation and publication in a peer-reviewed journal.

The RIST pilot and ensuing RCT will lead to improved management of wrist fractures and will address a gap in the current evidence base. The level 1 evidence generated from the definitive RCT will be published in peer-reviewed journals and presented at national and international meetings.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 55-70 and have had a distal radial fracture
2. The following radiographic findings before reduction: dorsal angulation ≤30 degrees, ulnar shortening ≤5 mm relative to the contralateral side (subjects will have contralateral wrist xrays), articular step ≤2 mm after initial post reduction and gap ≤5 mm

Exclusion Criteria:

1. patients with volarly displaced intra and extra articular fractures (Barton and Smith's)
2. radiocarpal subluxation or dislocation
3. open fractures
4. ipsilateral upper-extremity injuries
5. bilateral or multiple traumas

5) previous injury to the contralateral wrist

6) those deemed not suitable for surgical management (as indicated and documented by surgeon and research coordinator)

Ages: 55 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2015-05-22 (Actual); Primary Completion 2017-10-31 (Actual); Study Completion 2018-09-21 (Actual)

PRIMARY OUTCOMES:
Recruitment and eligibility rates | 1 year

SECONDARY OUTCOMES:
Patient Rated Wrist-Evaluation (PRWE) questionnaire | baseline, 6 weeks, 3 months, 6 months, and 12 months
Disabilities of the Arm, Shoulder, and Hand (DASH) Questionnaire | baseline, 6 weeks, 3 months, 6 months, 12 months
Visual Analogue Scale (VAS) for cosmesis | 6 weeks, 3 months, 6 months, 12 months
Visual Analogue Scale (VAS) for pain | baseline, 6 weeks, 3 months, 6 months, 12 months
Grip Strength (Hand held dynamometer) | baseline, 6 weeks, 3 months, 6 months, 12 months
Range of Motion (Goniometry) | baseline, 6 weeks, 3 months, 6 months, 12 months
Radiographic measures (Doral angulation, ulnar shortening, articular steps and gaps) | baseline, 6 weeks, 3 months, 6 months, 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Sturgeon Community Hospital, St. Albert, Alberta, Canada